CLINICAL TRIAL: NCT04382391
Title: A Prospective, Randomized, Controlled Study Assessing Vagus Nerve Stimulation in CoViD-19 Respiratory Symptoms (SAVIORII)
Brief Title: Study Assessing Vagus Nerve Stimulation in CoViD-19 Respiratory Symptoms
Acronym: SAVIORII
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A total of 21 patients were enrolled in the study resulting in 97 total collected specimen time points. Patient recruitment was halted due to greatly decreased numbers of patient hospitalizations for Covid-19.
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Collaborators: ElectroCore INC (Industry)
Responsible Party: Principal Investigator, Tariq Cheema, Associate Division Director, AHN Pulmonary, Critical Care and Sleep Medicine, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-132-AGH
Record Dates: First submitted 2020-04-14; First posted 2020-05-11 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: COVID; Corona Virus Infection; Respiratory Failure; Respiratory Distress Syndrome, Adult; ARDS, Human; SARS (Severe Acute Respiratory Syndrome)
MeSH Terms: conditions — Coronavirus Infections; Respiratory Insufficiency; Respiratory Distress Syndrome; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- gammaCore Sapphire® (nVNS) plus standard of care (Experimental): Subjects will be administered study treatment with the nVNS device 3 times per day (prophylaxis) and also as needed for acute respiratory symptoms.
  Interventions: Device: gammaCore® Sapphire (non-invasive vagus nerve stimulator); Other: Standard of care therapies
- standard of care alone (Active Comparator): Will receive standard of care therapies to treat CoViD-19 infection and symptoms
  Interventions: Other: Standard of care therapies

INTERVENTIONS:
Device: gammaCore® Sapphire (non-invasive vagus nerve stimulator) — Administer gammaCore® Sapphire daily, prophylactically, for three treatments (morning, mid-day and night, one hour before bed), each treatment consisting of two 2-minute doses/stimulations, one on each side of the neck. This would be a total of 6 treatments (2 doses x 3 times per day) of stimulation.
  For acute respiratory distress or shortness of breath (SOB), administer one treatment consisting of two 2-minute stimulations, on the neck. If respiratory distress or shortness of breath persists 20 minutes after the start of the first treatment, administer a second treatment.
  Arms: gammaCore Sapphire® (nVNS) plus standard of care
Other: Standard of care therapies — Will receive standard of care therapies for the treatment of CoViD-19 infection and symptoms

SUMMARY:
The study is a prospective, randomized, controlled investigation designed for comparison of two groups for the reduction of respiratory distress in a CoViD-19 population, using gammaCore Sapphire (nVNS) plus standard of care (active) vs. standard of care alone (SoC), the control group. The gammaCore® (nVNS) treatments will be used acutely and prophylactically. The aims of this study are to summarize and compare the incidence of clinical events and pro-inflammatory cytokine levels in patients randomized to use of gammaCore Sapphire plus standard of care vs standard of care alone in patients hospitalized for CoViD-19. Secondary objectives are demonstrate the safety of gammaCore Sapphire use in patients hospitalized for CoViD-19.

DETAILED DESCRIPTION:
Vagus nerve stimulation (VNS) has an established history of reducing airway distress. VNS has at least two mechanisms of action that may profoundly affect respiratory function in patients with respiratory distress due to CoViD-19.

First, vagus nerve stimulation modulates bronchoconstriction, acute stimulation has demonstrated a marked improvement in Work of Breathing (WOB) as well as Forced Expiratory Volume (FEV1) in patients with severe respiratory distress due to airway reactivity. This effect appears to occur via an afferent response to stimulation of the vagus nerve.

Second, and perhaps more importantly, VNS has been shown to be a potent moderator of pathologic immune reactions, specifically suppressing pro-inflammatory cytokine levels via activation of the Cholinergic Anti-inflammatory Pathway (CAP). VNS is currently being studied to modulate pro-inflammatory cytokines patterns and concentrations in a variety of acute and progressive inflammatory conditions, ranging from septic shock and asthma to stroke, rheumatoid arthritis and Inflammatory Bowel Disease. VNS has been studied in animal models of acute septic shock, consistently demonstrating life-saving potential. In one such study, cecal ligation and puncture was used to induce a septic state in an animal model. VNS reduced the expression of cytokines which was tightly associated with survival. Specifically, in animal and human models, this neuromodulatory therapy has the capacity to reduce the expression of inflammatory mediators, including TNF-α, IL-6 and IL-1β. These are precisely the same cytokines which are elevated in ARDS and other inflammatory disorders. In all cases, the therapy has shown considerable promise as a potential alternative to steroids (having potent anti-inflammatory activity but without the adverse side effects of steroids) and biologic therapies targeting pro-inflammatory cytokines (broadly - e.g., tofacitinib, or specifically - e.g., adalimumab, etanercept, and infliximab).

Viral-induced acute respiratory distress syndrome (ARDS), including those caused by SARS CoV-1 and MERS are characterized by a massive systemic pro-inflammatory state. Although a pro-inflammatory environment is required to control the rate of infection as well as the eradication of infected and compromised cells, the massive response to these viruses, primarily due to leukocytes of the innate arm of the immune system, is part of the problem as a significant number of tissues are damaged and lost secondary to the infected tissues in a by-stander and collateral manner. A simple, drug-free approach to attenuate this systemic inflammation would be of significant benefit to the progression of the syndrome and potentially improve the overall recovery of the patients.

For these reasons, the investigators propose that VNS may ameliorate the over-activity of the pro-inflammatory immune condition in CoViD-19 patients, thus conferring a superior therapeutic option especially for elderly patients and those presenting with respiratory illness in setting of co-morbid conditions who experience severe symptoms. These groups are at particularly high risk of requiring mechanical ventilation, developing ARDS, experiencing severe cytokine storm and have a higher mortality rate.

Non-Invasive Vagus Nerve Stimulation (nVNS) - Historically, VNS was delivered using implanted signal generators coupled to leads having electrodes that wrap around the vagus nerve. The vagus nerve is located within the carotid sheath, and thus the implantation surgery is complicated with inherent risks, particularly in the critically ill. More recently, a non-invasive approach to vagus nerve stimulation (nVNS) was cleared by the FDA for the acute treatment of pain associated episodic cluster and migraine headaches and the prevention of cluster headaches and migraine headaches. This device, gammaCore (electroCore, Inc., Basking Ridge, NJ) is handheld and requires no surgery or implants. The device is applied by healthcare providers or patients to the skin at the neck over the vagus nerve to deliver periodic doses of VNS non-invasively.

With respect to bronchoconstriction, early studies demonstrated modulation of airway reactivity in hospitalized asthmatic patients, improving various measures of airway patency.

Non-invasive VNS (nVNS) is a safe method of stimulating the vagus nerve, with minimal side effects. It does not require surgery or an invasive procedure that would otherwise limit its utility in the critically ill. The stimulation can be either self-administered or administered by a health care practitioner. There are numerous studies with both implanted and nVNS in multiple animal models and humans that have demonstrated a modulation of the inflammatory cascade with an improvement in survival.

gammaCore® (nVNS) has been studied in approximately 2,000 patients as part of clinical trials with an excellent safety profile. It is available through commercial insurers and the private pay market, and is listed on the federal supply schedule available for purchase by the VA and Department of Defense and also carries a CE mark for distribution abroad. More than ten thousand patients have been successfully treated in the United States and abroad.

CoViD-19 Respiratory Issues Involve Virally-triggered Severe (Lethal) Cytokine Expression - CoViD-19 (coronavirus disease 2019) is caused by SARS CoV-2 (severe acute respiratory syndrome coronavirus 2) and is related to the coronavirus which caused SARS in 2003 (SARS CoV-1). The virus is transmitted either through airborne droplets (e.g. coughing or sneezing) or direct contact (e.g. through a surface containing the virus), with a mean incubation period between 4 and 7 days (range 2 days to > 2 weeks). As of April 3, 2020, there are over a million confirmed cases and rising with 55,000 individuals deceased to date. This gives a current mortality rate of 5.3 %, although the base case of confirmed cases may be markedly underestimated. Elderly and those with co-morbid conditions including heart disease, diabetes, and asthma seem to have a higher mortality rate.

Many CoViD-19 patients experience moderate to severe respiratory symptoms, including shortness of breath and impaired oxygen saturation. Eighty-eight percent (88%) of patients present with respiratory symptoms. A significant and increasing number of CoViD-19 patients require hospitalization, and progress to being intubated and/or ventilator dependent. Given the rapid spread of this contagion, concern exists that the international healthcare systems do not have the number of ventilators and/or ICU beds to meet the expected demand in the coming months.

The most critically afflicted can experience pneumonia and/or ARDS. Accumulating evidence suggests that this subgroup with severe CoViD-19 likely have a cytokine storm syndrome, a hallmark of ARDS that includes dramatic increase in the expression of pro-inflammatory cytokines, mainly TNF-α, IL-6 and IL-1β among others. Elevations in IL-6 seem to be a particularly poor outcome indicator of respiratory compromise. It is believed that the mortality of ARDS is at least partially the result of an over activity of the patient's immune system.30 Predictors of fatality from a recent retrospective, multi-center study of 150 confirmed CoViD-19 cases in Wuhan, China, included elevated ferritin (mean 1297•6 ng/ml in non-survivors vs 614•0 ng/ml in survivors; p<0•001) and IL-6 (p<0•0001)31, suggesting that mortality and respiratory decompensation may be due to virally-driven hyperinflammation.

Therapies that could block the cytokine storm may help improve survival and decrease the need for ventilator use and prolonged respiratory support. Other companies are in fact developing pharmaceutical approaches for the treatment of cytokine storm, or plasma infusions from those who have recovered from the virus. At this point there is no cure or vaccine for the virus and neither is there a treatment approach to dampen the systemic inflammation.

Given the CE mark and excellent safety profile, including the twenty year history of the use of VNS to block the over production of pro-inflammatory mediators via the CAP (cholinergic anti-inflammatory pathway), and the lack of other effective or reasonable options during this pandemic the investigators propose deploying gammaCore® (nVNS) devices for prophylactic use to those who have been diagnosed as infected with the virus, but before the cytokine storm begins to cause and/or exacerbate the severe respiratory distress syndrome. The hypothesis is that the administration of non-invasive VNS using gammaCore®, during and following severe infection with CoViD-19 may prevent the worsening inflammatory response and acute injury associated, thus decreasing ventilator dependence and mortality of the virus. If utilized early enough in the course of disease the investigators hope to reduce ventilator dependence and improve survival with a scientifically driven safe and cost-effective approach. Furthermore, through additional acute utility of gammaCore® (nVNS) in cases of ARDS and cytokine storm the investigators can effectively blunt the pro inflammatory response, reduce mortality and liberate patients from mechanical ventilation earlier which will assist in deploying the ventilator to other patients in need during the CoViD-19 pandemic.

electroCore has designed a non-invasive vagus nerve stimulation (nVNS) device called gammaCore®. The gammaCore® (nVNS) device is a handheld, battery-powered unit that produces a proprietary electrical waveform in the vicinity of the vagus nerve in the neck. Each treatment, or dose, is relatively brief (120 seconds) and the user maintains control over the stimulation intensity.

gammaCore® is currently commercially available for the treatment of cluster and migraine headaches, and broad safety data with thousands of patients treated in the US Europe and the UK in both clinical trials and routine clinical care.

Treatment paradigms have been developed and tested in clinical trials to support FDA clearance for the acute treatment of pain associated with episodic cluster and migraine headaches, and the prevention of cluster and migraine headache. This experience demonstrates that nVNS may be administered safely in up to 24 two-minute doses per day. The investigators thus have data to draw on as to how to effectively stimulate the vagus nerve. Given the multiple modes of action with blocking the CAP, and acute bronchodilatation, using a similar treatment paradigm for a trial to evaluate nVNS treatment of ARDS is reasonable. The device should be used both prophylactically and acutely early in the course of the disease prior to mechanical ventilation, and once trained, treatment can be fully managed by either a healthcare professional or the patient. If one waits until mechanical ventilation has started, it is less likely that a therapy will be able to block the cytokine storm and outcomes will be less profound.

With respect to the theoretical cardiac and respiratory side effects of non-invasive treatment, historically, stimulation of the vagus nerve is associated with adverse side effects, including bradycardia and bronchoconstriction. These effects were shown to be the result of in discriminant stimulation of all fibers in the vagal bundle (the vagus nerve is primarily comprised of A and C fibers), which could be avoided by specifically tuning the electrical signals to selectively stimulate only the A fibers. This is possible because of the difference in electric field strengths necessary to activate the different fiber types.

The intensity, pulse duration and frequency of gammaCore® (nVNS) stimulation parameters have been optimized to induce signals in the large, myelinated Aβ fibers of the cervical branch of the vagus nerve. Since gammaCore® activates only the low threshold afferent Aβ fibers, versus the high threshold efferent C-fibers that innervate the heart, there is no known risk for adverse cardiac or other systemic parasympathetic effects.

electroCore has conducted pre-clinical studies to assess the potential risk of vagus nerve over-stimulation on the heart and airways. Several studies were conducted in beagle dogs with hypersensitized airways (worst case for airway reactivity) at maximum stimulation output for 2 minutes. Review of heart rate and airway resistance before, during and after stimulation indicated that there were no significant adverse changes associated with stimulation. These results are consistent with the human clinical experience with the gammaCore® device.

Regarding the theorized mechanism of action, afferent fibers from the vagus nerve enter the brain and synapse onto the nucleus tractus solitarius (NTS) in the brain stem , making connections with many structures in the brain including the locus coeruleus (LC), the periaqueductal gray (PAG) and the raphe nucleus (RN). These structures are known to control the release of key inhibitory neurotransmitters. Numerous animal and clinical studies over the last 25 years have implicated the activity of these structures, in particular the LC, in the mechanism of action of VNS to inhibit seizures.

Clinical Use for Clinical Care - Given the lack of other effective and/or reasonable options for a patient with CoViD-19 respiratory distress and the anticipated demands on our healthcare system, considering gammaCore® (nVNS) therapy, the investigators propose, is a reasonable approach. To achieve goal of decreasing health care burden with patient benefit of decreasing ventilator dependency, inflammatory response and mortality, plan to use it early in course of disease i.e. prior to severe respiratory distress and the need for mechanical ventilation.

The presumptive mechanisms of bronchodilatation and modulation of the cytokine storm would suggest that early intervention is ideal in improving pulmonary function and avoiding respiratory depression.

1. Prevention. Mitigation of pro-inflammatory immunokine release would be best achieved with two doses, consisting of a two-minute stimulation, on each side of the neck three times a day (am, afternoon and an hour before bed). This would be a total of 6 treatments (2 stimulations x 3 times per day) of stimulation as a prophylactic/preventive measure. This dosage is well below the known safety dosage threshold
2. In addition, patients may receive additional treatments when experiencing acute respiratory distress. Similarly, one treatment is two doses. Each treatment (a two-minute stimulation on each side of the neck) is performed on the neck. If shortness of breath (SOB) persists 20 minutes after start of first treatment, administer a second treatment. Maximum number of treatments per day is 9. This is symptomatic control and can be used to improve FEV1, Work of Breathing or dyspnea.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (age 18 years and older) who have tested positive or suspected/presumed positive for CoViD-19 using PCR real time test
2. Patients with cough, shortness of breath or respiratory compromise (RR>24/min, increased work of breathing.)
3. O2 Saturation less than or equal to 96% on room air or sensation
4. Agrees to use the gammaCore Sapphire device as intended and to follow all of the requirements of the study including recording required study data
5. Permission for early am blood draw to freeze for subsequent lab tests and sequencing as related to CoViD-19 sequelae
6. Patient is able to provide signed and witnessed Informed Consent

Exclusion Criteria:

1. On home/therapy oxygen (i.e. for chronic obstructive pulmonary disease (COPD) patients) at baseline prior to development of CoViD-19
2. Already using gammaCore® (nVNS) for other medical conditions
3. A history of aneurysm, intracranial hemorrhage, brain tumors, or significant head trauma
4. Known or suspected severe atherosclerotic cardiovascular disease, severe carotid artery disease (e.g., bruits or history of transient ischemic attack or cerebrovascular accident), congestive heart failure, known severe coronary artery disease, myocardial infarction documented within past 90 days, or current or recent history of life-threatening arrhythmia (sustained ventricular tachycardia, ventricular fibrillation, second or third-degree heart block, uncontrolled atrial fibrillation or uncontrolled atrial flutter)
5. Patients with clinically significant hypertension, hypotension, bradycardia, or tachycardia (as per investigator discretion)
6. Current implantation of an electrical and/or neurostimulator device, including but not limited to a cardiac pacemaker or defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant
7. Current implantation of metal cervical spine hardware or a metallic implant near the gammaCore® stimulation site
8. Belongs to a vulnerable population or has any condition such that his or her ability to provide informed consent, comply with the follow-up requirements, or provide self-assessments is compromised (e.g. homeless, developmentally disabled and prisoner)
9. Compromised access to peripheral veins for blood sampling.
10. Pregnant women
11. Patients with active cancer or those who have had recent cancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2023-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Cheema, MD, Principal Investigator — Allegheny Health Network; Boyle Cheng, PhD, Study Director — Allegheny Health Network
Locations (2):
- United States (2):
  - AHN Allegheny General Hospital, Pittsburgh, Pennsylvania
  - AHN West Penn Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 patients enrolled into the study: 11 control patients, 10 experimental (nVNS arm); First patient consented on 15May2020 and final patient consented on 09Feb2021. Original enrollment target was 60 patients, however, enrollment slowed as number of inpatient Covid cases decreased, thus creating it difficult to enroll. New and approved treatment options became available for this population, thus it was determined to close enrollment in this trial prior to achieving 60 patients.
Groups:
- gammaCore Sapphire® (nVNS) Plus Standard of Care: Subjects will be administered study treatment with the nVNS device 3 times per day (prophylaxis) and also as needed for acute respiratory symptoms.
  gammaCore® Sapphire (non-invasive vagus nerve stimulator): Administer gammaCore® Sapphire daily, prophylactically, for three treatments (morning, mid-day and night, one hour before bed), each treatment consisting of two 2-minute doses/stimulations, one on each side of the neck. This would be a total of 6 treatments (2 doses x 3 times per day) of stimulation.
  For acute respiratory distress or shortness of breath (SOB), administer one treatment consisting of two 2-minute stimulations, on the neck. If respiratory distress or shortness of breath persists 20 minutes after the start of the first treatment, administer a second treatment.
  Standard of care therapies: Will receive standard of care therapies for the treatment of CoViD-19 infection and symptoms
Period: Overall Study
Arm/Group | gammaCore Sapphire® (nVNS) Plus Standard of Care | Standard of Care Alone
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | gammaCore Sapphire® (nVNS) Plus Standard of Care | Standard of Care Alone | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 6 | 9 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21
Requiring Intubation [Count of Participants; unit: Participants] | 0 | 0 | 0
mean oxygen saturation (baseline) [Mean (Full Range); unit: Percent saturation of peripheral oxygen] | 91.6 [80 to 98] | 92.8 [83 to 97] | 92.2 [80 to 98]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Events
Description: compare clinical events between the control group and active group for patients admitted to the hospital for CoViD-19.
Time Frame: From baseline to 90 days post-discharge
Measure: Count of Participants; unit: Participants
Arm/Group | gammaCore Sapphire® (nVNS) Plus Standard of Care | Standard of Care Alone
Number analyzed (Participants) | 10 | 11
Participants
  Number of participants with SAE | 5 | 5
  Number of participants intubated while hospitalized for COVID-19 | 1 | 1
  Death up to 90 days post-discharge | 0 | 1

2. Secondary Outcome: Evaluate C-reactive Protein (CRP) Trends
Description: measure the changes in the serum/plasma concentrations of CRP
Time Frame: From baseline to discharge from hospital or death while hospitalized (patients had data for up to 6.2 days on average after baseline for these outcomes)
Measure: Mean (Full Range); unit: milligrams per deciliter
Arm/Group | gammaCore Sapphire® (nVNS) Plus Standard of Care | Standard of Care Alone
Number analyzed (Participants) | 10 | 11
milligrams per deciliter
  CRP baseline | 13.7 [0 to 34] | 7.7 [1.3 to 14.2]
  CRP Peak | 17.4 [0 to 39.3] | 14 [1.9 to 42.5]
  CRP at discharge or death | 2.6 [0 to 7.9] | 5.1 [0 to 36.9]

3. Secondary Outcome: Evaluate Supplemental Oxygen Requirements
Description: compare the difference in oxygen requirements (liters/min) between the control group and active group for patients admitted to the hospital for CoViD-19.
Time Frame: as for outcome 2
Measure: Mean (Full Range); unit: fraction of inspired oxygen (percentage)
Arm/Group | gammaCore Sapphire® (nVNS) Plus Standard of Care | Standard of Care Alone
Number analyzed (Participants) | 10 | 11
fraction of inspired oxygen (percentage)
  highest FiO2 requirement while hospitalized | 54.4 [28 to 100] | 57.3 [21 to 100]
  FiO2 requirement at discharge | 29.2 [21 to 52] | 30.8 [21 to 100]

4. Secondary Outcome: Number of Participant Deaths
Description: number of participant deaths due to Covid-19
Time Frame: as for outcome 2
Measure: Number; unit: number of deaths
Arm/Group | gammaCore Sapphire® (nVNS) Plus Standard of Care | Standard of Care Alone
Number analyzed (Participants) | 10 | 11
number of deaths | 0 | 1

5. Secondary Outcome: Time to Onset of Mechanical Ventilation
Description: Time to mechanical ventilation between control group and treatment group (for patients who progress to the need for mechanical ventilation)
Time Frame: From baseline to discharge from hospital or death while hospitalized
Population: Note that only one patient in each group required mechanical ventilation.
Measure: Number; unit: days
Arm/Group | gammaCore Sapphire® (nVNS) Plus Standard of Care | Standard of Care Alone
Number analyzed (Participants) | 1 | 1
days | 9.0 | 15.3

6. Secondary Outcome: Compare Clinical Improvement in Participants
Description: World Health Organization (WHO) Ordinal Scale for Clinical Improvement.
Time Frame: From baseline to discharge from hospital or death while hospitalized (data not collected during the study for this outcome)
Population: incomplete sample size due to early termination, did not collect WHO data for analysis
Arm/Group | gammaCore Sapphire® (nVNS) Plus Standard of Care | Standard of Care Alone
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Evaluate Ferritin Levels/Trends
Description: measure the changes in the serum/plasma concentrations of Ferritin
Time Frame: as for outcome 2
Measure: Mean (Full Range); unit: nanograms per mililiter
Arm/Group | gammaCore Sapphire® (nVNS) Plus Standard of Care | Standard of Care Alone
Number analyzed (Participants) | 10 | 11
nanograms per mililiter
  Ferritin baseline | 915.6 [87 to 2209] | 762.9 [54 to 2903]
  Ferritin Peak | 1256.6 [178.6 to 3307] | 1463.9 [205 to 6655]
  Ferritin at discharge or death | 704.2 [136.7 to 1858] | 1124.9 [67 to 6655]

8. Secondary Outcome: Evaluate D-dimer Trends/Levels
Description: measure the changes in the serum/plasma concentrations of D-Dimer
Time Frame: as for outcome 2
Measure: Mean (Full Range); unit: mcg per mL fibrinogen equivalent unit
Arm/Group | gammaCore Sapphire® (nVNS) Plus Standard of Care | Standard of Care Alone
Number analyzed (Participants) | 10 | 11
mcg per mL fibrinogen equivalent unit
  D-Dimer baseline | 5.0 [0.8 to 14.1] | 1.0 [0.4 to 1.9]
  D-Dimer Peak | 7.9 [1 to 19.1] | 3.7 [1 to 20]
  D-Dimer at discharge or death | 1.8 [0.4 to 10.5] | 2.2 [0.4 to 13.2]

9. Secondary Outcome: Evaluate Pro-Calcitonin (PCT) Levels/Trends
Description: measure the changes in the serum/plasma concentrations of Pro-Calcitonin
Time Frame: as for outcome 2
Population: 1 participant in the treatment arm did not have Pro-Calcitonin drawn at any timepoints; 1 participant in control arm did not have discharge Pro-calcitonin drawn
Measure: Mean (Full Range); unit: nanograms per mililiter
Arm/Group | gammaCore Sapphire® (nVNS) Plus Standard of Care | Standard of Care Alone
Number analyzed (Participants) | 10 | 11
nanograms per mililiter
  Pro-Calcitonin baseline: number analyzed (Participants) | 9 | 11
  Pro-Calcitonin baseline | 2.9 [0.06 to 23.8] | 0.2 [0.08 to 0.54]
  Pro-Calcitonin Peak: number analyzed (Participants) | 9 | 11
  Pro-Calcitonin Peak | 2.9 [0.06 to 23.8] | 1.1 [0.08 to 9.84]
  Pro-Calcitonin at discharge or death: number analyzed (Participants) | 9 | 10
  Pro-Calcitonin at discharge or death | 0.1 [0.04 to 0.32] | 1.0 [0.04 to 9.84]

10. Secondary Outcome: Evaluate Cytokine Trends (Serum/Plasma Level of TNF-α)
Description: The level of the cytokine TNF-α in serum/plasma, as measured using ELISA.
Time Frame: From baseline up to 7 days, discharge or death (whichever occurred first)
Population: The analysis population was determined for study day 0, 1, 2, 3, 5 and 7 based on how many patients were still enrolled in the study on that day and had cytokine data that could be evaluated.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | gammaCore Sapphire® (nVNS) Plus Standard of Care | Standard of Care Alone
Number analyzed (Participants) | 10 | 11
pg/mL
  Day 0 | 17.1 (23.1) | 77.9 (164.7)
  Day 1: number analyzed (Participants) | 9 | 11
  Day 1 | 14.2 (17.4) | 89.7 (175.8)
  Day 2: number analyzed (Participants) | 8 | 7
  Day 2 | 14.8 (16.8) | 83.5 (183.1)
  Day 3: number analyzed (Participants) | 7 | 8
  Day 3 | 21.6 (40.1) | 60.0 (136.2)
  Day 5: number analyzed (Participants) | 4 | 5
  Day 5 | 20.6 (31.6) | 73.9 (132.2)
  Day 7: number analyzed (Participants) | 1 | 5
  Day 7 | 0.0 (NA) — Standard deviation cannot be calculated because only one patient in this group had data for Day 7 | 15.6 (14.4)

11. Secondary Outcome: Evaluate Cytokine Trends (Serum/Plasma Level of IL-1β)
Description: The level of the cytokine IL-1β in serum/plasma, as measured using ELISA.
Time Frame: From baseline up to 7 days, discharge or death (whichever occurred first)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | gammaCore Sapphire® (nVNS) Plus Standard of Care | Standard of Care Alone
Number analyzed (Participants) | 10 | 11
pg/mL
  Day 0 | 3.7 (6.2) | 47.3 (83.5)
  Day 1: number analyzed (Participants) | 9 | 11
  Day 1 | 4.4 (7.3) | 53.4 (98.8)
  Day 2: number analyzed (Participants) | 8 | 7
  Day 2 | 4.6 (6.6) | 48.3 (91.6)
  Day 3: number analyzed (Participants) | 7 | 8
  Day 3 | 5.9 (9.0) | 42.9 (86.8)
  Day 5: number analyzed (Participants) | 4 | 5
  Day 5 | 2.2 (3.8) | 65.1 (105.5)
  Day 7: number analyzed (Participants) | 1 | 5
  Day 7 | 0.0 (NA) — Standard deviation cannot be calculated because only one patient in this group had data for Day 7 | 17.3 (26.9)

12. Secondary Outcome: Evaluate Cytokine Trends (Serum/Plasma Level of IL-6)
Description: The level of the cytokine IL-6 in serum/plasma, as measured using ELISA.
Time Frame: From baseline up to 7 days, discharge or death (whichever occurred first)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | gammaCore Sapphire® (nVNS) Plus Standard of Care | Standard of Care Alone
Number analyzed (Participants) | 10 | 11
pg/mL
  Day 0 | 101.7 (129.2) | 68.9 (66.7)
  Day 1: number analyzed (Participants) | 9 | 11
  Day 1 | 58.7 (89.7) | 74.7 (65.0)
  Day 2: number analyzed (Participants) | 8 | 7
  Day 2 | 82.9 (141.0) | 63.3 (54.5)
  Day 3: number analyzed (Participants) | 7 | 8
  Day 3 | 60.8 (92.9) | 69.0 (64.4)
  Day 5: number analyzed (Participants) | 4 | 5
  Day 5 | 114.7 (167.6) | 60.8 (65.3)
  Day 7: number analyzed (Participants) | 1 | 5
  Day 7 | 0.0 (NA) — Standard deviation cannot be calculated because only one patient in this group had data for Day 7 | 35.3 (20.5)

ADVERSE EVENTS:
Time Frame: up to 3 months post discharge, an average of 3.5 months
Arm/Group | gammaCore Sapphire® (nVNS) Plus Standard of Care | Standard of Care Alone
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/11
Serious Adverse Events (participants affected / at risk) | 5/10 | 5/11
Other Adverse Events (participants affected / at risk) | 2/10 | 2/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | gammaCore Sapphire® (nVNS) Plus Standard of Care (N=10) | Standard of Care Alone (N=11)
Pleuritic chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
critical illness myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
bacteremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
deep vein thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
tracheostomy (Surgical and medical procedures) | 1 (1) | 0 (0)
severe malnutrition (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urachal diverticulum infection (Infections and infestations) | 1 (1) | 0 (0)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
hypertension (Cardiac disorders) | 0 (0) | 1 (1)
intubation (Surgical and medical procedures) | 1 (1) | 1 (1)
anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
exertional hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | gammaCore Sapphire® (nVNS) Plus Standard of Care (N=10) | Standard of Care Alone (N=11)
fatigue (General disorders) | 1 (1) | 1 (1)
hypertension (Cardiac disorders) | 1 (1) | 0 (0)
tachycardia (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment slowed as number of inpatient Covid cases decreased and the number of experimental therapies increased, thus creating it difficult to enroll. New and approved treatment options became available for this population, thus it was determined to close enrollment in this trial prior to meeting enrollment goal. Early termination lead to smaller number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT04382391/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT04382391/ICF_002.pdf